CLINICAL TRIAL: NCT03774303
Title: Effectiveness of Mobile Application Intervention on Preschool Children's Fear and Pain and Their Parents' Anxiety and Stress in Day Surgery
Brief Title: Effectiveness of Mobile Application Intervention in Day Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HAK
Record Dates: First submitted 2018-11-27; First posted 2018-12-12 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Pain; Fear; Stress; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile intervention (Experimental): families to be prepared for day surgery with a mobile application
  Interventions: Other: Mobile application
- control group (Active Comparator): families to be prepared for day surgery with current practice
  Interventions: Other: current practice

INTERVENTIONS:
Other: Mobile application — A mobile application that will be used to prepare families for day surgery
  Arms: mobile intervention
Other: current practice — the current practice used to prepare families for day surgery
  Arms: control group

SUMMARY:
In Finland about 50% of surgical operations for all under 16 years of age are made as day surgery which means that the patient comes to the hospital and is discharged on the day of the operation. Day surgery will continue to grow in the next few years. Its benefits include shorter hospitalization, family reunion and rapid recovery. The preschool children and their parents who come in for day surgery feel fear, anxiety and stress, which depend on the amount of knowledge and its quality. By developing the preparation of preschool children and their parents for day surgery, and by testing new methods more attention can be paid to the special features of day surgery, supporting the families, and increasing family involvement in the whole process.

The purpose of this study is to describe and evaluate the effectiveness of a new mobile application intervention compared to the effectiveness of the traditional preparing method when measuring preschool children's fear and pain and their parents' anxiety and stress. The aim is to produce new information and to develop day surgery of preschool children.

The study consist of two phases. The first phase of the research is a systematic literature review and meta-analysis. The purpose of the review is to assess and describe the methods previously used in the preparation of parental day surgery and their effectiveness for preschool children fear and pain and parents' anxiety and stress. The second phase of the study is carried out as a randomized controlled trial (=RCT). The parents of the preschool children are randomized to the mobile application group (n = 50-60) and the control group (n = 50-60). The sample size is based on power-analysis, with anxiety as the primary outcome. The material for the second phase of the study is collected at the day surgery department of the Oulu University Hospital. The study group is prepared for day surgery with a new mobile application and the control group according to the traditional preparing method. The study examines the effectiveness of a new intervention compared to the effectiveness of the traditional preparing method when measuring preschool children's fear and pain and their parents' anxiety and stress. The collected data are analyzed using the Mann-Whitney, t-test, Khi square test, and Fisher's accurate test.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or 2
* ELECTIVE DAY SURGIGAL PROCEDURE IN 3-4 WEEKS
* PARENT ABLE TO USE MOBILE INTERVENTION, UNDERSTANDS FINNISH AND WILLING TO PARTICIPATE IN PREPARING CHILD FOR DAY SURGERY
* GENERAL ANAESTHESIA

Exclusion Criteria:

* INCLUSION CRITERIA NOT MET

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Parents' Anxiety measured with STAI-Y1. | first measurement at home before the procedure
  The STAI meter is a two-part adult anxiety meter developed by Charles D. Spielberg and his research team (1983). It separates situation related anxiety (STATE-A = Y1) from character related tendency towards anxiety (TRAIT-A). In this study, the most commonly used version of the STAI meter and only it's STATE-A section is utilized. Here, the parent evaluates his own current anxiety on a four-step scale with twenty questions. The respondents choose from the following options at each question: 1 = no anxiety at all, 2 = slight anxiety, 3 = some anxiety 4 = very much anxiety.
Parents' Anxiety measured with STAI-Y1. | second measurement in the hospital before the procedure
  The STAI meter is a two-part adult anxiety meter developed by Charles D. Spielberg and his research team (1983). It separates situation related anxiety (STATE-A = Y1) from character related tendency towards anxiety (TRAIT-A). In this study, the most commonly used version of the STAI meter and only it's STATE-A section is utilized. Here, the parent evaluates his own current anxiety on a four-step scale with twenty questions. The respondents choose from the following options at each question: 1 = no anxiety at all, 2 = slight anxiety, 3 = some anxiety 4 = very much anxiety.
Parents' Anxiety measured with STAI-Y1. | third measurement in the hospital before discharge
  The STAI meter is a two-part adult anxiety meter developed by Charles D. Spielberg and his research team (1983). It separates situation related anxiety (STATE-A = Y1) from character related tendency towards anxiety (TRAIT-A). In this study, the most commonly used version of the STAI meter and only it's STATE-A section is utilized. Here, the parent evaluates his own current anxiety on a four-step scale with twenty questions. The respondents choose from the following options at each question: 1 = no anxiety at all, 2 = slight anxiety, 3 = some anxiety 4 = very much anxiety.
Parents' Anxiety measured with STAI-Y1. | fourth measurement at home within 1-7 days after the procedure
  The STAI meter is a two-part adult anxiety meter developed by Charles D. Spielberg and his research team (1983). It separates situation related anxiety (STATE-A = Y1) from character related tendency towards anxiety (TRAIT-A). In this study, the most commonly used version of the STAI meter and only it's STATE-A section is utilized. Here, the parent evaluates his own current anxiety on a four-step scale with twenty questions. The respondents choose from the following options at each question: 1 = no anxiety at all, 2 = slight anxiety, 3 = some anxiety 4 = very much anxiety.

SECONDARY OUTCOMES:
Parents' Stress with VRSS | first measurement at home before the procedure
  VRSS (short Verbal Rating Scale for Stress). The VRSS meter measures stress experienced by the parent. The meter consists of six claims: 0 = I did not feel stress at all 1 = I felt little stress 2 = I felt some stress 3 = I felt quite a lot of stress 4 = I felt a lot of stress 5 = I felt the worst stress imaginable.
Parents' Stress with VRSS | second measurement in the hospital before the procedure
  VRSS (short Verbal Rating Scale for Stress). The VRSS meter measures stress experienced by the parent. The meter consists of six claims: 0 = I did not feel stress at all 1 = I felt little stress 2 = I felt some stress 3 = I felt quite a lot of stress 4 = I felt a lot of stress 5 = I felt the worst stress imaginable.
Parents' Stress with VRSS | third measurement in the hospital before discharge
  VRSS (short Verbal Rating Scale for Stress). The VRSS meter measures stress experienced by the parent. The meter consists of six claims: 0 = I did not feel stress at all 1 = I felt little stress 2 = I felt some stress 3 = I felt quite a lot of stress 4 = I felt a lot of stress 5 = I felt the worst stress imaginable.
Parents' Stress with VRSS | fourth measurement at home within 1-7 days after the procedure
  VRSS (short Verbal Rating Scale for Stress). The VRSS meter measures stress experienced by the parent. The meter consists of six claims: 0 = I did not feel stress at all 1 = I felt little stress 2 = I felt some stress 3 = I felt quite a lot of stress 4 = I felt a lot of stress 5 = I felt the worst stress imaginable.
Children's Fear with FAS | first measurement at home before the procedure
  FAS (Facial Affective Scale). The FAS meter measures the child's fear with nine facial images and describes its intensity ranging from no fear to the worst possible fear.
Children's Fear with FAS | second measurement in the hospital before the procedure
  FAS (Facial Affective Scale). The FAS meter measures the child's fear with nine facial images and describes its intensity ranging from no fear to the worst possible fear.
Children's Fear with FAS | third measurement in the hospital before discharge
  FAS (Facial Affective Scale). The FAS meter measures the child's fear with nine facial images and describes its intensity ranging from no fear to the worst possible fear.
Children's Fear with FAS | fourth measurement at home within 1-7 days after the procedure
  FAS (Facial Affective Scale). The FAS meter measures the child's fear with nine facial images and describes its intensity ranging from no fear to the worst possible fear.
Children's Pain with PPPM | first measurement at home before the procedure
  PPPM (Parent's Postoperative Pain Measure). The PPPM meter measures pain behavior of children aged 1 to 6 years of age as assessed by their parents. The PPPM meter is divided into a section for 1-to 2 -year-old children and another section for 3- to 6 -year-olds.
Children's Pain with PPPM | second measurement in the hospital before the procedure
  PPPM (Parent's Postoperative Pain Measure). The PPPM meter measures pain behavior of children aged 1 to 6 years of age as assessed by their parents. The PPPM meter is divided into a section for 1-to 2 -year-old children and another section for 3- to 6 -year-olds.
Children's Pain with PPPM | third measurement in the hospital before discharge
  PPPM (Parent's Postoperative Pain Measure). The PPPM meter measures pain behavior of children aged 1 to 6 years of age as assessed by their parents. The PPPM meter is divided into a section for 1-to 2 -year-old children and another section for 3- to 6 -year-olds.
Children's Pain with PPPM | fourth measurement at home within 1-7 days after the procedure
  PPPM (Parent's Postoperative Pain Measure). The PPPM meter measures pain behavior of children aged 1 to 6 years of age as assessed by their parents. The PPPM meter is divided into a section for 1-to 2 -year-old children and another section for 3- to 6 -year-olds.
Children's Pain with VAS | first measurement at home before the procedure
  VAS (Visual Analogy Scale). The VAS scale allows the parents to evaluate the intensity of the pain of their children on a 10cm long scale that starts at zero meaning no pain at all and ends at 10 representing the worst possible pain. Preschool children evaluate their pain with a face scale, also where zero means no pain and ten means the worst possible pain.
Children's Pain with VAS | second measurement in the hospital before the procedure
  VAS (Visual Analogy Scale). The VAS scale allows the parents to evaluate the intensity of the pain of their children on a 10cm long scale that starts at zero meaning no pain at all and ends at 10 representing the worst possible pain. Preschool children evaluate their pain with a face scale, also where zero means no pain and ten means the worst possible pain.
Children's Pain with VAS | third measurement in the hospital before discharge
  VAS (Visual Analogy Scale). The VAS scale allows the parents to evaluate the intensity of the pain of their children on a 10cm long scale that starts at zero meaning no pain at all and ends at 10 representing the worst possible pain. Preschool children evaluate their pain with a face scale, also where zero means no pain and ten means the worst possible pain.
Children's Pain with VAS | fourth measurement at home within 1-7 days after the procedure
  VAS (Visual Analogy Scale). The VAS scale allows the parents to evaluate the intensity of the pain of their children on a 10cm long scale that starts at zero meaning no pain at all and ends at 10 representing the worst possible pain. Preschool children evaluate their pain with a face scale, also where zero means no pain and ten means the worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerimaa H, Polkki T. Effectiveness of Digital Counseling for Parents' Use of Nonpharmacological Pain-Relieving Methods in Pediatric Day Surgery. Pain Manag Nurs. 2025 Oct;26(5):544-554. doi: 10.1016/j.pmn.2025.04.011. Epub 2025 May 22. PMID 40410077
- [Derived] Kerimaa H, Hakala M, Haapea M, Vahanikkila H, Serlo W, He HG, Polkki T. Effectiveness of a Mobile App Intervention for Preparing Preschool Children and Parents for Day Surgery: Randomized Controlled Trial. J Med Internet Res. 2023 Sep 29;25:e46989. doi: 10.2196/46989. PMID 37773624